CLINICAL TRIAL: NCT06225908
Title: The Effects of Serratus Posterior Superior Intercostal Plane Block on Postoperative Analgesia in Patients Undergoing Breast Cancer Surgery
Brief Title: SPSIPB for Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Bengü Gülhan Köksal, Principal Investigator, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-12-13/12
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Pain, Postoperative; Pain, Acute; Opioid Consumption
Keywords: breast surgery; pain management
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Control (No Intervention)
- Group SPSİPB (Active Comparator)
  Interventions: Procedure: Serratus posterior superior intercostal plane block

INTERVENTIONS:
Procedure: Serratus posterior superior intercostal plane block — application of local anestesic under serratus posterior superior muscle at the level of second costa
  Arms: Group SPSİPB

SUMMARY:
Acute postoperative pain after breast cancer surgery is usually moderate to severe, and inadequate postoperative pain management can significantly increase perioperative analgesic consumption, prolong hospital stay, and even cause long-term persistent pain such as postmastectomy pain syndrome. A multimodal analgesic approach (NSAII, paracetamol, opioids, local infiltration, facial plane blocks and paravertebral and periparavertebral blocks) is recommended.

Paravertebral block (PVB) is considered the gold standard analgesic method for breast surgery. However, PVB is an invasive block requiring advanced skills and deep injection in close proximity to the pleura, intercostal nerves, neuraxis, great vessels and intercostal neurovascular bundles. As a result, the ongoing risks of pneumothorax, neuraxial spread, hypotension and systemic toxicity preclude its routine use in the day surgery setting. Therefore, alternative blocks have been developed. Various regional techniques such as Serratus plan block (SPB), interpectoral/pectoroserratus blocks (PECS I/II), erector spina plan block (ESPB) and rhomboid intercostal plan block (RIB) have been used to relieve pain after breast surgery. However, local anesthetic distribution may be affected by the surgical incision in the chest muscles. ESPB can be performed from cervical to sacral vertebrae, but clinical, cadaveric and radiologic results are inconsistent. RIB provides hemithoracic analgesia; however, RIB does not cover the cranial aspect of the T2 dermatome. A meta-analysis reported that SPB effectively relieves acute postoperative pain, reduces nausea and vomiting, and improves perioperative anesthesia outcomes in breast surgery. In another study compared with placebo, it was reported that serratus plane block provided less pain at rest, but there was no significant difference in reducing postoperative opioid consumption.

Serratus Posterior Superior Intercostal Plan Block is performed in the fascial plane between the serratus posterior superior muscle and intercostal muscles at the second and third costal level. SPSIB provides hemithoracic analgesia from the paraspinal region to the anteromedial region of the chest wall including the axillary region. In a case series of patients undergoing breast surgery, it was reported that the costal plane plays an important role in preventing pneumothorax, provides a natural barrier to the pleura, and may be a good choice for postoperative analgesia management as part of multimodal analgesia after breast surgery.

In this study, the investigators aimed to observationally investigate the effect of serratus posterior superior intercostal plane block on postoperative opioid consumption in patients undergoing breast cancer surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* ASA I-II-III risk group
* Patients whose consent was obtained with an informed consent form
* Breast Cancer Surgery operation patients who will undergo

Exclusion Criteria:

* Under 18 and over 65
* ASA ≥ IV
* History of allergy to local anesthetics
* Known coagulation disorders
* Infection near the entry site
* Chronic use of analgesics
* Diabetes Mellitus and patients receiving neoadjuvant chemotherapy
* Body Mass index over 30
* Dementia or confusion
* Lack of cooperation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
opioid consumption | up to 24 hour after surgery
  total consumption of opioid during 24 hour after surgery

SECONDARY OUTCOMES:
Pain scores | up to 24 hour after surgery
  Patient's pain intensity by using numeric rating scale score

CONTACTS AND LOCATIONS:
Locations (1):
- Zongulak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koksal BG, Baytar C, Bayraktar E, Balbaloglu H. Effects of serratus posterior superior intercostal plane block on postoperative analgesia in patients undergoing breast cancer surgery: a randomized controlled trial. BMC Anesthesiol. 2025 Apr 24;25(1):209. doi: 10.1186/s12871-025-03092-0. PMID 40275145